CLINICAL TRIAL: NCT01326338
Title: Multi-Center, Double-Blind, Placebo-Controlled Study of Nitazoxanide Suspension in the Treatment of Prolonged Diarrhea in Children
Brief Title: Nitazoxanide for the Treatment of Prolonged Diarrhea in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Celine Rossignol, MS, Romark Laboratories, L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM02-3019
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Diarrhea
Keywords: Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitazoxanide Suspension (Experimental): Nitazoxanide Oral Suspension 100 mg/5 ml for patients aged 1-3 years or Nitazoxanide Oral Suspension 200 mg/10 ml for patients aged 4-11 years
  Interventions: Drug: Nitazoxanide
- Placebo Suspension (Placebo Comparator): Placebo Oral Suspension 5 ml for patients aged 1-3 years and Placebo Oral Suspension 10 ml for patients aged 4-11 years
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide Oral Suspension 100 mg/5 ml for patients aged 1-3 years twice daily for 3 days or Nitazoxanide Oral Suspension 200 mg/10 ml for patients aged 4-11 years twice daily for 3 days
  Other Names: Alinia

SUMMARY:
The purpose of this study was to determine the efficacy of nitazoxanide suspension compared to placebo in treating prolonged diarrhea in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diarrhea ≥3 days but <30 days duration.
* No visible blood in stool.

Exclusion Criteria:

* Use of any antibacterial, antiparasitic or antiviral drugs within 5 days of enrollment.
* Females who are pregnant, suspected of being pregnant or breastfeeding.
* Serious systemic disorders incompatible with the study.
* History of hypersensitivity to nitazoxanide.
* Patients in whom the possibility of receiving placebo and not being able to receive immediately an effective treatment will be incompatible with the severity of the patient's illness according to the investigator's judgment.
* Patients known to have or suspected of having AIDS or other immune deficiencies.

Ages: 12 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2005-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Time from first dose to resolution of symptoms | Up to 17 days
  Resolution of symptoms defined as resolution of all gastrointestinal symptoms associated with prolonged diarrhea at enrollment including abdominal pain or tenderness, distention, etc. with the patient not requiring anti-motility or other palliative treatment. Symptom resolution must be maintained for at least 72 hours to be considered valid.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Lopez, MD, Principal Investigator — Regional Hospital of Cajamarca
Locations (1):
- Regional Hospital of Cajamarca, Cajamarca, Peru

REFERENCES:
- [Derived] Rossignol JF, Lopez-Chegne N, Julcamoro LM, Carrion ME, Bardin MC. Nitazoxanide for the empiric treatment of pediatric infectious diarrhea. Trans R Soc Trop Med Hyg. 2012 Mar;106(3):167-73. doi: 10.1016/j.trstmh.2011.11.007. Epub 2012 Jan 31. PMID 22301075